CLINICAL TRIAL: NCT07209241
Title: Phase Ib, Open-Label Study of CART-EGFR-IL13Rα2 Cells Administered Following Lymphodepleting Chemotherapy or Prior to Surgical Resection in Patients With EGFR-Amplified Recurrent Glioblastoma
Brief Title: Different Approaches for CART-EGFR-IL13Ra2 Dosing in Recurrent GBM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10325
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: This study will evaluate three different approaches for administering CART-EGFR-IL13Ra2 cells in the setting of recurrent glioblastoma. Each dosing approach will be evaluated as a separate treatment arm as outlined below:
  * Arm A: Single Fixed-Dose Administration Following Lymphodepletion
  * Arm B: Repeat Dose Administration Following Lymphodepletion
  * Arm C: Single Fixed-Dose Administration in the Pre-Operative Setting
  Subjects are assigned sequentially, beginning with Arm A. Once Arm A is fully enrolled and all safety evaluations are complete, the data, along with cumulative data from other CART-EGFR-IL13Ra2 studies, will be reviewed by the Clinical Principal Investigator (PI) and Sponsor Medical Director to determine whether to open Arm B.
  If it is decided not to progress to Arm B for any reason, Arm A will be expanded to include up to a total of eight evaluable subjects. Enrollment into Arm C begins only after Arms A and B (if applicable) are fully enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): Subjects will receive a single fixed-dose administration of CART-EGFR-IL13Ra2 cells following lymphodepletion.
  Interventions: Biological: CART-EGFR-IL13Ra2 T cells
- Arm B (Active Comparator): Subjects will receive repeated dose administration of CART-EGFR-IL13Ra2 cells following lymphodepletion.
  Interventions: Biological: CART-EGFR-IL13Ra2 T cells
- Arm C (Active Comparator): Subjects will receive a single fixed-dose administration of CART-EGFR-IL13Ra2 in the pre-operative setting.
  Interventions: Biological: CART-EGFR-IL13Ra2 T cells

INTERVENTIONS:
Biological: CART-EGFR-IL13Ra2 T cells — CART-EGFR-IL13Ra2 cells are autologous T cells co-expressing two CARs targeting the cryptic EGFR epitope 806 and IL13Ra2.

SUMMARY:
This is an open-label, phase 1b study to evaluate different approaches for CART-EGFR-IL13Ra2 dosing and further characterize the safety, feasibility, preliminary efficacy, and pharmacokinetics of CART-EGFR-IL13Ra2 cells in patients with EGFR-amplified glioblastoma that has recurred following prior radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written informed consent
2. Male or female age ≥ 18 years
3. Patients with glioblastoma, IDH-wildtype (as defined by WHO 2021 Classification of CNS Tumors) that has recurred following prior radiotherapy1. For patients with tumors harboring methylation of the MGMT promoter, a t l east 1 2 w eeks must have elapsed since completion of first-line radiotherapy.
4. Tumor tissue positive for wild-type EGFR amplification by NeoGenomics Laboratories. Archival tumor from patient's initial surgery at time of original diagnosis or recently collected tumor from time of recurrence are acceptable.
5. Surgical tumor resection for disease control/management (Arms A, B, C) or tumor biopsy to confirm tumor recurrence (Arms A and B only) is clinically indicated in the opinion of the physician-investigator.
6. Adequate organ function defined as:

   1. Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 30 ml/min and not on dialysis.
   2. ALT/AST ≤ 3 x ULN
   3. Total bilirubin ≤ 2.0 mg/dL, except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome (≤ 3.0 mg/dL)
   4. Left Ventricular Ejection Fraction (LVEF) ≥ 45% confirmed by ECHO/MUGA
   5. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air
7. Karnofsky Performance Status ≥ 60%.
8. Subjects of reproductive potential must agree to use acceptable birth control methods, as described in protocol Section 4.3.

Exclusion Criteria:

1. Active hepatitis B or hepatitis C infection.
2. Any other active, uncontrolled infection.
3. Class III/IV cardiovascular disability according to the New York Heart Association Classification
4. Tumors primarily localized to the brain stem or spinal cord.
5. Severe, active co-morbidity in the opinion of the physician-investigator that would preclude participation in this study.
6. Receipt of bevacizumab within 3 months prior to physician-investigator confirmation of eligibility.
7. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10 mg daily of prednisone. Patients with autoimmune neurological diseases (such as MS or Parkinson's) will be excluded.
8. Patients who are pregnant or nursing (lactating).
9. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2042-11-01 (Estimated); Study Completion 2042-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with treatment related adverse events using NCI Common Terminology Criteria for Adverse Events (CTCAE) V5.0 | Up to 15 years following CART-EGFR-IL13Ra2 administration
  Type, frequency, severity, and attribution of adverse events
Occurrence of treatment-limiting toxicities (Arms A and B only) | Up to 28 days following CART-EGFR-IL13Ra2 administration
  Type, frequency, severity, and attribution of treatment limiting adverse events as defined in protocol section 8.1.7

SECONDARY OUTCOMES:
Evaluate the feasibility of different approaches for CART-EGFR-IL13Ra2 dosing | Up to 2 years
  Proportion of eligible subjects who receive study treatment.
  Proportion of eligible subjects assigned to arm B who receive all planned doses of CART-EGFR-IL13Ra2 cells
Progression-free Survival (PFS) | Up to 15 years following CART-EGFR-IL13Ra2 administration
  Per RANO 2.0 criteria
Overall Survival (OS) | Up to 15 years following CART-EGFR-IL13Ra2 administration
  Per RANO 2.0 criteria
Objective Response Rate (ORR) | Up to 15 years following CART-EGFR-IL13Ra2 administration
  Per RANO 2.0 criteria in participants with measurable disease at the time of study treatment (Treatment Arms A and B) or Post-Surgical Resection (Treatment Arm C)
Duration of response (DOR) | Up to 15 years following CART-EGFR-IL13Ra2 administration
  Per RANO 2.0 criteria in participants with measurable disease at the time of study treatment (Treatment Arms A and B) or Post-Surgical Resection (Treatment Arm C)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bagley, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States